CLINICAL TRIAL: NCT02496338
Title: Effect of Menopausal Health Training for Husbands on Women's Quality of Life and Marital Satisfaction During Transitional Period
Brief Title: Menopausal Health Training for Husbands on Women's Quality of Life and Marital Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gonabad University of Medical Sciences (Other)
Collaborators: Shahid Sadoughi University of Medical Sciences and Health Services (Other)
Responsible Party: Principal Investigator, Narjes Bahri, Faculty Member in Department of Midwifery, Gonabad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 92/11
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Menopause
Keywords: Menopause; Quality of Life; Marital Satisfaction; training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Training program about menopausal health isues
  Interventions: Other: Training program about menopausal health isues
- Control group (No Intervention): No training program about menopausal health isues

INTERVENTIONS:
Other: Training program about menopausal health isues — A three sessions raining program about health issues during menopause for spouses of 45-60 years old
  Arms: Intervention group

SUMMARY:
The investigators conducted a clinical trial to evaluation the effect of a menopausal health training for Husbands of 45-60 years women on the women's quality of life and marital satisfaction during transitional period to menopause.

DETAILED DESCRIPTION:
The investigators applied a menopausal health training program for Husbands of 45-60 years women. The content of menopausal health training program was about the nature of menopause, signs and symptoms, complications, treatment option and health behavior during transitional period. Training program lasted 3 sessions. The investigators assessed quality of life and marital satisfaction using Hildich marital satisfaction questionnaire and Menopause Quality of Life questionnaire(MENQOL), respectively, three month after intervention.

ELIGIBILITY:
Inclusion Criteria:

* living with their spouse
* no history of premature menopause
* no history of hysterectomy
* no history of oophorectomy
* no history of acute disease
* no history of burden chronic disease

Exclusion Criteria:

* no participation of spouse in all of training session
* uncompleted all of equation
* favorite to exclude from study

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 3 months
  assessing with MENQOL

SECONDARY OUTCOMES:
Marital satisfaction | 3 months
  Hildich Marital satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: MahamadAli MorovvatiSharifabad, PhD, Study Chair — Yazd University of Medical Sicences